CLINICAL TRIAL: NCT01718288
Title: Optimization of Treatment in Patients With Severe Peripheral Ischemia (Fontaine Stage IIb), Unsuitable or Suitable to Surgical Revascularization / Endovascular With Reference to the Change of Pain-free Walking Distance and Other Endpoints
Brief Title: Optimization of Treatment in Patients With Severe Peripheral Ischemia (Fontaine Stage IIb)
Acronym: 2bPILOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eudract Number: 2006-001660-23
Record Dates: First submitted 2012-10-22; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; iloprost; walking distance; cardiovascular events
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Iloprost; Aspirin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- iloprost + standard treat.(aspirin) (Experimental): 1B - patients unsuitable to surgical or endovascular vascular therapy: treatment with iloprost intravenous infusions for 10 days every 3 months, in addition to conventional treatment
  Interventions: Drug: iloprost; Drug: Standard Treatment (aspirin.....),
- Standard Treatment (aspirin....) (Active Comparator): 1A - patients unsuitable to surgical or endovascular vascular therapy: conventional treatment
  Conventional Treatments:correction of concomitant risk factors, physical exercise, antiplatelet, standard heparin / low molecular weight heparin, hemorheological / vasodilators such as pentoxifylline / buflomedil, propionyl-L-carnitine, Defibrotide) but not prostanoids
  Interventions: Drug: Standard Treatment (aspirin.....),
- Vascular surgery patients + iloprost (Experimental): 2B - patients suitable to vascular surgical or endovascular therapy: treatment with intravenous infusions iloprost for 10 days every 3 months, in addition to conventional treatment
  Interventions: Drug: iloprost; Drug: Standard Treatment (aspirin.....),
- Vasc. Surg.+ standard treat. (aspirin..) (Active Comparator): 2A - patients suitable to vascular surgical or endovascular therapy + standard treatment (aspirin...)
  Interventions: Drug: Standard Treatment (aspirin.....),

INTERVENTIONS:
Drug: iloprost — The study, consists of two substudies, which deal with patients susceptible to medical therapy alone (substudy 1) or treated with classical surgical therapy (substudy 2).
  For each substudy, pts will be divided into two groups, one that will receive conventional treatments but not prostanoids, other conventional treatments with addition of iloprost.
  The 4 groups:
  1A. Pts unsuitable to surgical or endovascular vascular therapy: conventional treatment
  1. B. Pts unsuitable to surgical or endovascular vascular therapy: treatment with iloprost plus conventional treatment
  2. A. Pts suitable to vascular surgical or endovascular therapy: conventional treatment
  2B. Pts suitable to vascular surgical or endovascular therapy: treatment with iloprost plus conventional treatment
  Other Names: ENDOPROST*0,05MG/0,5ML 1F
  Arms: Vascular surgery patients + iloprost; iloprost + standard treat.(aspirin)
Drug: Standard Treatment (aspirin.....), — The standard treatment, as has already been explained in the submission is the best treatment that the guidelines suggest for that specific type of patient with those complications and with stage 2b severe PAD.
  correction of concomitant risk factors, physical exercise, antiplatelet, standard heparin /low molecular weight heparin, hemorheological/vasodilators such as pentoxifylline/buflomedil, propionyl-L-carnitine, Defibrotide) but not prostanoids
  Other Names: aspirin, antiplatelet, statins,hemorheological/vasodilators

SUMMARY:
Evaluate the possibility of optimization of therapy with prostanoids (iloprost), in patients with Fontaine's stage IIb severe chronic ischemia, both in patients eligible for surgery both in patients for which it is only possible medical therapy

DETAILED DESCRIPTION:
The management of patients with peripheral arterial disease (PAD) stage IIb and pain-free walking distance (PFWD) less than 100 meters is a major clinical problem, in view of the significant cooling of the quality of life and evolution often severe that characterizes the clinical course of these patients. Revascularization Surgery is the treatment of choice, but about half of patients with severe PAD IIb is not eligible for surgery or endovascular treatment. The usefulness of use of vasodilators or hemorheological is controversial, and medical treatment of these patients is therefore heterogeneous understanding the various pharmacologic options (for the correction of risk factors, prevention of cardiovascular events, improvement of claudication), and rehabilitative programs. Iloprost, a synthetic analogue of prostacyclin, is effective in the treatment of patients with chronic critical ischemia, and its pharmacological profile (effective vasodilator, anti-platelet, and leukocyte activation) is particularly suitable to modulate multiple components pathogenesis of peripheral arterial disease. Specifically, in the treatment of patients with PAD IIb severe, the current state is available only a retrospective study that compared the use of iloprost with that of vasodilators. Aim of the study FADOI-2bPILOT is to evaluate prospectively and for an observation period of 13 months, if you can get a benefit on the pain-free walking distance and on clinical outcome from "anticipated" and additional use of iloprost, in patients with severe IIb stage PAD treated according to current "best medical practice".

ELIGIBILITY:
Inclusion Criteria: age > 18 years; pain-free walking distance (PFWD) <100 meters on two occasions 10 days apart, with <25% difference between each other; ankle blood pressure (BP) <70 mmHg; big toe BP < 30 mmHg (in case of diabetic patient).

Exclusion Criteria: pain at rest, trophic ulcers or gangrene (critical limb ischemia), if they were unable to cooperate, or one of the following conditions (contraindications or precautions for use of iloprost) was present: myocardial infarction or stroke in the previous 6 months; congestive heart failure NYHA class >II; unstable angina; uncontrolled severe arterial hypertension (systolic BP >180 mmHg or diastolic BP >110 mmHg) or hypotension (systolic BP <90 mmHg); hyperkinetic ventricular arrhythmia; acute pulmonary edema or pulmonary congestion; bleeding diathesis; platelet count <80,000 or > 500,000/mm3; renal failure requiring dialysis; liver cirrhosis; pregnancy or breast feeding; history of allergy, hypersensitivity or intolerance to iloprost or other prostanoids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-11; Primary Completion 2011-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Measure of PFWD(pain-free walking distance)in patients with 2b stage PAD | 13 months
  Aim of this multicenter, randomized, controlled study was prospectively evaluate the effects of iloprost, added to standard therapy, in patients with 2b stage PAD and PFWD (pain-free walking distance) less than 100 metres, eligible and non-eligible for surgical revascularization. A treadmill test 3-6-9-12 months (before iloprost cycle for patients group 1B and 2B). A final evaluation 13 months (for one month to the conclusion of the 12 months treatment of iloprost for patients group 1B and 2B, and after 13 months from enrolling for patients in the study group 1A and 2A)

SECONDARY OUTCOMES:
Assessing changes in endurance | 13 months
  A clinical evaluation 3-6-9-12 months (before iloprost cycle for patients group 1B and 2B). A final evaluation 13 months (for one month to the conclusion of the 12 months treatment of iloprost for patients group 1B and 2B, and after 13 months from enrolling for patients in the study group 1A and 2A)
The possible occurrence of major complications | 13 months
  The study reported the number of events during all the study (13 months). The major complication were: Ischemic cardiopathy, critical limb ischemia, cerebrovascular event, critical limb ischemia
Quality of life | 13 months
  For the Quality of life, the study used a specific questionnaire administrated to all patients enrolled in the study (13 months of observation): IQOLA (International Quality of Life Assessment),SF-36 Italian Version 1.6

CONTACTS AND LOCATIONS:
Overall Officials: Gualberto Gussoni, MD, PhD, Study Director — Fadoi Foundation
Locations (14):
- Italy (14):
  - Angiology, Hospital "G. Fucito", Mercato San Severino, Salerno
  - Internal Medicine, Hospital "Policlinico", Bari
  - Angiology, Hospital "Ferrarotto - Alessi", Catania
  - Internal Medicine, Hospital "Pugliese - Ciaccio", Catanzaro
  - Internal Medicine, Hospital of Fermo, Fermo
  - Vascular Surgery, Hospital "Galliera", Genoa
  - Internal Medicine, Hospital Civile, Legnano
  - Internal Medicine, "Madonna delle Grazie" Hospital, Matera
  - Internal Medicine, Hospital "Fatebenefratelli", Naples
  - Surgery Dept., Hospital " San Giovanni Bosco", Naples
  - Internal Medicine, Hospital "Bianchi Melacrino Morelli", Reggio Calabria
  - Internal Medicine, Hospital Policlinico Campus Biomedico, Rome
  - Internal Medicine, Hospital "Fondazione Circolo Macchi", Varese
  - Internal Medicine, Hospital "Jazzolino", Vibo Valentia